CLINICAL TRIAL: NCT03125525
Title: Clinical Experience With Transcutaneous Supraorbital Nerve Stimulation in Patients With Refractory Migraine or With Migraine and Intolerance to Topiramate: a Prospective Exploratory Clinical Study
Brief Title: Clinical Experience With Transcutaneous Supraorbital Nerve Stimulation in Refractory Migraine
Status: Completed | Type: Observational
Sponsor: Corfu Headache Clinic (Other)
Responsible Party: Principal Investigator, KONSTANTINOS SPINGOS, Dr., Corfu Headache Clinic
Other Study IDs: CorfuHC
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Migraine
Keywords: migraine; transcutaneous; supraorbital; nerve; stimulation
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Active treatment patients: Patients using Cefaly device on routine daily basis
  Interventions: Device: Cefaly device

INTERVENTIONS:
Device: Cefaly device — Use of Cefaly based upon the protocol of the approval study of the device, in which it is used once every day on the migraine prevention program
  Other Names: transcutaneous supraorbital nerve stimulation with Cefaly

SUMMARY:
Migraine is included in the top-ten disabling diseases and conditions among the Western populations. Non-invasive neurostimulation (t-SMS), including the Cefaly® device, for the treatment of various types of pain is a relatively new field of interest. The aim of the present study was to explore the clinical experience with Cefaly® in a cohort of migraine patients previously refractory or non-tolerant to topiramate prophylaxis.

Patients were followed prospectively after having been diagnosed with episodic or chronic migraine with a previous failure to topiramate treatment and having consented to receive preventive treatment with Cefaly® according to their treating physician's suggestion. A 1-month period of baseline observation was followed by a 3-month period of active treatment with transcutaneous supraorbital nerve stimulation (t-SNS) with Cefaly® as the only preventive treatment.

DETAILED DESCRIPTION:
Migraine is ranked as the sixth most disabling condition, worldwide.Presently, medications are the mainstream of migraine management; however, preventive treatment is often far from optimal. Preventive treatment for migraine is usually considered when migraine pain is present more frequently than twice a week.

Topiramate is currently the most commonly used first-line approved preventive medication for migraine. With this being said, not all patients respond to preventive medications, due to either lack of efficacy or to adverse events. As a matter of fact, adherence to migraine preventive medications, including topiramate, may be insufficient. In a health insurance database based review, 70.2% of patients who initiated migraine prophylaxis with antiepileptics were reported to be non-adherent after 6 months. Among preventive medication choices, patients are reported to adhere best, but not optimally to topiramate, with adverse events being the most common reason for topiramate discontinuation.

On the other hand, non-invasive neurostimulation is a relatively new field of interest for the treatment of various types of pain. Clinical research in this field is active, as the recent technological advances allow for safe, convenient and ease by which to self-administer treatment sessions. Cefaly® electrically the supraorbital nerve in the forehead. The supraorbital nerve is a branch of the first trigeminal division. The trigeminovascular system has a well-known involvement in headache pain. Transcutaneous supraorbital nerve stimulation (t-SNS) with the Cefaly® (Cefaly® Technology sprl, Herstal, Belgium) device has proved to be a safe and efficient method for convenient self-delivered treatment sessions. It has received approval for the prevention of episodic migraine by the American Food and Drug Administration and by the EU, including Greece, since early 2015.

Although t-SNS use is spreading in Greece, it is not reimbursed by the social security system and in many cases it may be postponed until either a first line preventive medication fails to provide substantial relief or tolerability / safety issues ensue.

The aim of the present study was to explore and share the clinical experience with Cefaly® in a cohort of migraine patients previously refractory or intolerant to preventive treatment with topiramate, as this is a common situation in clinical practice. Additionally, we specifically explored whether the reason for the discontinuation of topiramate is correlated with the outcome of Cefaly® treatment. To the best of the authors' knowledge, no similar study has been published so far.

METHODS This was an exploratory prospective multicenter clinical study conducted in accordance with the principles of the Helsinki Declaration and approved by the principal investigator's (MV) Institutional Review Board. This study was done to explore the efficiency and safety of Cefaly® in migraine prevention in a population of patients previously refractory or intolerant to topiramate.

Participants to be treated with Cefaly® were enrolled from 2 private headache clinics, located in Athens and Thessaloniki, the first and second largest cities of Greece, respectively. Patients were diagnosed with episodic or chronic migraine, needed preventive treatment according to the treating physician's opinion, and they had not responded to previous topiramate treatment, either due to inefficacy or due to intolerability or safety issues. In order to consider topiramate as failed due to inefficacy, a dose of 100mg/day for at least 3 months was required to have been received. Topiramate was considered as failed due to intolerability in any case a patient had decided to stop use of topiramate due to an adverse event regardless of its nature or severity. Patients had to have stopped topiramate at least 3 months prior to starting treatment with Cefaly®.

Both episodic and chronic (≥ 15 days of headache per month) migraine patients, according to the International Classification of Headache Disorders 3rd edition-beta version (ICHD IIIβ), were included. Upon enrolment and after giving consent to participate in the study, demographics and clinical data were captured, including the reason for topiramate discontinuation. Patients were then provided with a headache (HA) diary to be self-completed over the course of the study including questions about occurrence of HA, peak intensity level on a 0-10 numerical scale, number of acute medication doses and any adverse event. A 1-month baseline observation period was followed by a 3-month active treatment period with Cefaly® as the only preventive treatment. During the active treatment period, compliance (days the device was used as recommended, e.g. 1 full session each day) was also recorded.

The European version of Cefaly® includes three stimulation programs; one for acute migraine relief and two programs to be implemented in daily 20-minute sessions, one for migraine prevention and one for relaxation. In our study, Cefaly® was to be used based upon the protocol of the approval study of the device, in which it is used once every day on the migraine prevention program.

At their last evaluation, patients answered two additional questions regarding their total subjective satisfaction from treatment with t-SNS. The first question ("Are you satisfied with Cefaly® and wish to continue the treatment?") was aimed to access overall satisfaction from t-SNS treatment and the will to continue treatment, which was the primary evaluation of our study. The second question ("Did you encounter technical issues with the device?") was aimed to access any problems or technical difficulties arising from the use of the device.

Changes in total headache days, number of HA days with intensity ≥5/10 and days with acute medication use were analysed from baseline to the last observation or Month-3 of active treatment.

ELIGIBILITY:
Inclusion Criteria:

- Migraine according to the criteria of International Headache Society classification III lack of response or intolerance to topiramate. Patient's consent

Exclusion Criteria:

- No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients non-respondint to preventive treatment of migraine with topiramate accepting to use Cefaly according to protocol proposed by their treating phycisian
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change in headache days | 4 months
  Change in headache days, as recorded on a self-administered headache questionnaire, at 1st, 2nd and 3rd month of active treatment comparing to the baseline observation.
  Linear Mixed Models were performed, with patients modelled as a random effect, time (study month), and their interaction modelled as fixed effects.
  Statistical significance was set to the observed level of 5%. All statistical analyses were performed using STATA v.13.

SECONDARY OUTCOMES:
Patient overall satisfaction | 3 months
  Patients resonse to the question "Are you satisfied with Cefaly® and wish to continue the treatment?"

CONTACTS AND LOCATIONS:
Overall Officials: Michail Vikelis, Study Director — Meditteraneo Hospital of Athens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Riederer F, Penning S, Schoenen J. Transcutaneous Supraorbital Nerve Stimulation (t-SNS) with the Cefaly(R) Device for Migraine Prevention: A Review of the Available Data. Pain Ther. 2015 Oct 14;4(2):135-47. doi: 10.1007/s40122-015-0039-5. Online ahead of print. PMID 26467451
- [Derived] Vikelis M, Dermitzakis EV, Spingos KC, Vasiliadis GG, Vlachos GS, Kararizou E. Clinical experience with transcutaneous supraorbital nerve stimulation in patients with refractory migraine or with migraine and intolerance to topiramate: a prospective exploratory clinical study. BMC Neurol. 2017 May 18;17(1):97. doi: 10.1186/s12883-017-0869-3. PMID 28521762
- See also: Cefaly® Technology. (Last accessed 27 Jul. 16) — http://www.cefalytechnology.com/en/company